CLINICAL TRIAL: NCT05428176
Title: Leveraging Digital Health Solutions to Reduce Learning and Functional Disparities in Children With Cancer
Brief Title: A High Intensity Electronic Health Intervention for the Reduction of Learning Disparities in Childhood Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22057; NCI-2022-04695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22057 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Neuropsychologists blinded to arm assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (high intensity e-Health program) (Experimental): Patients and parents receive the high intensity eHealth intervention through the interactive website and via videoconferencing for 30-50 minutes once every 3 to 4 weeks for up to 5 sessions over 6 months. Patients and parents also receive usual care. After 6 months, parents attend booster sessions at months 7, 9, and 11.
  Interventions: Other: Best Practice; Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients and parents receive usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
Other: Internet-Based Intervention — Undergo eHealth intervention
  Arms: Arm I (high intensity e-Health program)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a high intensity electronic health (eHealth) intervention program for reducing learning disparities in children with cancer. Most children with leukemia and lymphoblastic lymphoma can be cured due to advancements in diagnosis and treatment. However, because treatments for these conditions target the central nervous system, these children are at increased risk for developing neurocognitive late effects (problems with attention, thinking, learning, and remembering). Fortunately, many survivors do well, but some children continue to struggle with learning and have academic difficulties after their cancer treatments. The purpose of this research study is to see whether providing parents with educational knowledge and parenting tips using videoconferencing and a special website better helps their cancer survivor child in learning and school achievement compared to typical services.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effectiveness of high intensity program (HIP)-eHealth on pediatric cancer survivors' learning and school-related outcomes up to 12 months post-enrollment.

SECONDARY OBJECTIVES:

I. Determine the effectiveness of HIP-eHealth on parental efficacy up to 12 months post-enrollment.

II. Examine the extent to which parents' self-reported efficacy and/or children's use of online learning activities correlates with the children's school functioning.

III. Examine differences in HIP-eHealth uptake and effects across socio-demographic groups.

OUTLINE:

PRE-STUDY: Parent-child dyads attend 4 intervention sessions over 10 weeks and provide feedback in support of intervention refinement.

Parent-child dyads are randomized to 1 of 2 arms.

ARM I: Patients and parents undergo high intensity eHealth intervention through the interactive website and via videoconferencing for 30-50 minutes once every 3 to 4 weeks for up to 5 sessions over 6 months. Patients and parents also receive usual care. After 6 months, parents attend booster sessions at months 7, 9, and 11.

ARM II: Patients and parents receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Primary participating parent/caregiver is English- or Spanish-speaking (any race/ethnicity)
* Child is aged 6-12 years (yr.) (for the website usability pre-study, child is age 8 - 12 yrs.)
* Child understands English (but can be bilingual)
* Child treated for acute leukemia (e.g., acute lymphoblastic leukemia, acute myelogenous leukemia) or lymphoblastic lymphoma
* Child is in cancer remission and has completed cancer therapies, including maintenance treatment
* Primary participating parent/caregiver has daily contact with the child
* Child is enrolled in school

Exclusion Criteria:

* Recent or current participation in a behavioral intervention study with a similar focus
* History of major psychiatric condition (e.g., psychosis) in parent or child
* Severe neurodevelopmental disorder in the child (e.g., down syndrome, intellectual disability)
* Child has previously used the IXL online learning program extensively and unwilling to regularly use it again
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Child's improvement in academic functioning | At baseline and 1 year
  Measured using the Wechsler Individual Achievement Test (WIAT) Numerical Operations (NO) subset. The WIAT NO score at 1 year will be compared between treatment arms using the Generalized Estimating Equation (GEE), adjusting for baseline values and accounting for correlations among patients within a study site. An indicator variable for treatment arm will be included in the model, its significance tested, and a 95% confidence interval constructed.

SECONDARY OUTCOMES:
Objective academic performance (Child) | Up to 5 years
  Assessed by WIAT reading and math scores, grades from school report cards, IXL diagnostic scores in math and English language arts (high intensity program e-health group only). The GEE will also be used to compare the effects of high intensity program e-Health intervention and low intensity program on this outcome. Non-normally distributed measurements will be transformed to achieve normality. If this is not possible, they will be dichotomized, and GEE for binary outcomes will be used for analysis. Potential modification of the treatment effect by covariates (e.g., child's age, parent's language, sex/gender, race/ethnicity, time since diagnosis) will be explored by including the two-way interaction of treatment by covariate. Will also perform subgroup analysis by estimating the within-subgroup intervention effects and constructing the 95% confidence intervals in groups defined by the covariates, e.g. sex/gender (men, women) and language (English, Spanish).
Attention performance (Child) | Up to 5 years
  Assessed with Conners Parent Report Attention and Hyperactivity subscales. The GEE will also be used to compare the effects of high intensity program e-Health intervention and low intensity program on this outcome. Non-normally distributed measurements will be transformed to achieve normality. If this is not possible, they will be dichotomized, and GEE for binary outcomes will be used for analysis. Potential modification of the treatment effect by covariates (e.g., child's age, parent's language, sex/gender, race/ethnicity, time since diagnosis) will be explored by including the two-way interaction of treatment by covariate. Will also perform subgroup analysis by estimating the within-subgroup intervention effects and constructing the 95% confidence intervals in groups defined by the covariates, e.g. sex/gender (men, women) and language (English, Spanish).
Parent-reported functioning of child (Child) | Up to 5 years
  Assessed by Pediatric Quality of Life Inventory Psychosocial Functioning: School, Emotional, Social domains. The GEE will also be used to compare the effects of high intensity program e-Health intervention and low intensity program on this outcome. Non-normally distributed measurements will be transformed to achieve normality. If this is not possible, they will be dichotomized, and GEE for binary outcomes will be used for analysis. Potential modification of the treatment effect by covariates (e.g., child's age, parent's language, sex/gender, race/ethnicity, time since diagnosis) will be explored by including the two-way interaction of treatment by covariate. Will also perform subgroup analysis by estimating the within-subgroup intervention effects and constructing the 95% confidence intervals in groups defined by the covariates, e.g. sex/gender (men, women) and language (English, Spanish).
Use of learning strategies (Child) | Up to 5 years
  Assessed with School Motivation and Learning Strategies Inventory study strategies subscale, student self-regulatory strategy use scale. The GEE will also be used to compare the effects of high intensity program e-Health intervention and low intensity program on this outcome. Non-normally distributed measurements will be transformed to achieve normality. If this is not possible, they will be dichotomized, and GEE for binary outcomes will be used for analysis. Potential modification of the treatment effect by covariates (e.g., child's age, parent's language, sex/gender, race/ethnicity, time since diagnosis) will be explored by including the two-way interaction of treatment by covariate. Will also perform subgroup analysis by estimating the within-subgroup intervention effects and constructing the 95% confidence intervals in groups defined by the covariates, e.g. sex/gender (men, women) and language (English, Spanish).
Mean of item scores from the Student Intrinsic Motivation to Learn questionnaire | Baseline, time 2, time 3
  Student Intrinsic Motivation to Learn Questionnaire measuring motivation for academic learning
Mean of item scores from the Student Academic Self-efficacy questionnaire | Baseline, time 2, time 3
  .Student Academic Self-efficacy measures self-confidence
Knowledge of pro-learning parenting (Parents) | Up to 5 years
  Assessed with Parent Beliefs and Behaviors Questionnaire (PBQ-R3) knowledge scale. GEE models using one indicator variable of time will be used to examine the efficacy of the high intensity program eHealth intervention compared to low intensity program on these scores, adjusting for baseline measurements and study site, and accounting for within-site and within-individual correlations. Other parent-related covariates that are imbalanced at baseline will be included in the model. The efficacy of the intervention will be assessed by testing the significance of the interaction of treatment-by-time indicator.
Frequency of pro-learning behaviors (Parents) | Up to 5 years
  Assessed with PBQ-R3 parenting behaviors scale, and weekly time spent with the child in pro-learning behaviors and activities. GEE models using one indicator variable of time will be used to examine the efficacy of the high intensity program eHealth intervention compared to low intensity program on these scores, adjusting for baseline measurements and study site, and accounting for within-site and within-individual correlations. Other parent-related covariates that are imbalanced at baseline will be included in the model. The efficacy of the intervention will be assessed by testing the significance of the interaction of treatment-by-time indicator.
Parenting pro-learning efficacy (Parents) | At baseline, 6 months, 1 year
  Assessed with PBQ-R3 efficacy scale. GEE models using one indicator variable of time will be used to examine the efficacy of the high intensity program eHealth intervention compared to low intensity program on these scores, adjusting for baseline measurements and study site, and accounting for within-site and within-individual correlations. Other parent-related covariates that are imbalanced at baseline will be included in the model. The efficacy of the intervention will be assessed by testing the significance of the interaction of treatment-by-time indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Sunita K Patel, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of Calif San Francisco, San Francisco, California